CLINICAL TRIAL: NCT06490003
Title: Predicting Postoperative Chemotherapy Efficacy in Patients With Esophageal Squamous Cell Carcinoma by Biopsy Specimens.
Brief Title: Predicting Postoperative Chemotherapy Efficacy in Patients With Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/ESCC-Chemo
Record Dates: First submitted 2024-06-21; First posted 2024-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemotherapy Effect; DNA Methylation
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Fluorouracil; Cisplatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Formalin-fixed and paraffin-embedded (FFPE) samples derived from biopsy specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy response patients.: Responders according to the response evaluation criteria in solid tumors (RECIST).
  A panel of DNA methylation, whose specific methylation level is tested DNA from resection tissue with Methylation-specific PCR(MSP)
  Interventions: Drug: Fluoro Uracil
- Chemotherapy non-response patients: Responders according to the response evaluation criteria in solid tumors (RECIST).
  A panel of DNA methylation, whose specific methylation level is tested DNA from resection tissue with Methylation-specific PCR(MSP)
  Interventions: Drug: Fluoro Uracil

INTERVENTIONS:
Drug: Fluoro Uracil — Esophageal cancer chemotherapy（First line treatment)
  Other Names: Cisplatin

SUMMARY:
Esophageal cancer remains a disease with a poor prognosis. Chemotherapy is an important part of its treatment, but there are cases in which chemotherapy is ineffective. The investigators aim to develop a model to predict the response to chemotherapy by DNA methylation of preoperative biopsy specimens to identify the chemotherapy ineffective group.

DETAILED DESCRIPTION:
Esophageal cancer remains a disease with a poor prognosis. In the treatment of esophageal squamous cell carcinoma (ESCC), multidisciplinary treatment including surgery, chemotherapy, and radiation therapy is important. Chemotherapy is an effective treatment for esophageal cancer, but some patients do not respond to it. Non-response to chemotherapy can result in disease progression, loss of patient fitness, and even the opportunity to receive other treatments that might have originally had a therapeutic effect. If there are biomarkers that could indicate the efficacy of chemotherapy before treatment, ineffective patients would be able to change their treatment plan. Patients on preoperative chemotherapy would be able to avoid unnecessary chemotherapy and undergo surgery without the effects of physical weakness and side effects. On the other hand, patients on definitive chemotherapy may choose to intensify their treatment with additional radiation therapy or immunotherapy. The investigators aim to develop a model to predict the response to chemotherapy by DNA methylation of preoperative biopsy specimens to identify the chemotherapy ineffective

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had histologically confirmed esophageal squamous cell carcinoma.
2. Patients who had undergone chemotherapy.
3. Patients receiving initial chemotherapy
4. Written informed consent following full study information is provided to the patient.

Exclusion Criteria:

1. Patients for whom a preoperative biopsy sample cannot be obtained
2. Patients who cannot assess at 2 months later after chemotherapy.
3. Patients with multiple cancers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chemotherapy naive patient needed esophageal squamous cell carcinoma chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2004-06-01 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(Chemotherapy) | 1year
  The effect of initial chemotherapy is evaluated by imaging. Response evaluation criteria in solid tumors (RECIST) is used for treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Takiguchi, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- Yamanashi Universiy, Chūō, Yamanashi, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Morgan E, Soerjomataram I, Rumgay H, Coleman HG, Thrift AP, Vignat J, Laversanne M, Ferlay J, Arnold M. The Global Landscape of Esophageal Squamous Cell Carcinoma and Esophageal Adenocarcinoma Incidence and Mortality in 2020 and Projections to 2040: New Estimates From GLOBOCAN 2020. Gastroenterology. 2022 Sep;163(3):649-658.e2. doi: 10.1053/j.gastro.2022.05.054. Epub 2022 Jun 4. PMID 35671803
- [Background] Shah MA, Kennedy EB, Catenacci DV, Deighton DC, Goodman KA, Malhotra NK, Willett C, Stiles B, Sharma P, Tang L, Wijnhoven BPL, Hofstetter WL. Treatment of Locally Advanced Esophageal Carcinoma: ASCO Guideline. J Clin Oncol. 2020 Aug 10;38(23):2677-2694. doi: 10.1200/JCO.20.00866. Epub 2020 Jun 22. PMID 32568633
- [Background] Macedo-Silva C, Constancio V, Miranda-Goncalves V, Leite-Silva P, Salta S, Lobo J, Guimaraes R, Carvalho-Maia C, Gigliano D, Farinha M, Sousa O, Henrique R, Jeronimo C. DNA methylation biomarkers accurately detect esophageal cancer prior and post neoadjuvant chemoradiation. Cancer Med. 2023 Apr;12(7):8777-8788. doi: 10.1002/cam4.5623. Epub 2023 Jan 20. PMID 36670548
- [Background] Zhang Y, Cao Y, Zhang J, Huang M, Roy P, Huang B, Yang H, Rong Y, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Lin J, Zhang J, Fu J, He J, Li H. Lymph Node Ratio Improves Prediction of Overall Survival in Esophageal Cancer Patients Receiving Neoadjuvant Chemoradiotherapy: A National Cancer Database Analysis. Ann Surg. 2023 Jun 1;277(6):e1239-e1246. doi: 10.1097/SLA.0000000000005450. Epub 2022 Jul 6. PMID 35797545
- [Background] Zhang XY, Yan WP, Sun Y, Li XT, Chen Y, Fan MY, Wu Y, Liang Z, Xiong HC, Wang ZL, Sun YS, Chen KN. CT Signs Can Predict Treatment Response and Long-Term Survival: A Study in Locally Advanced Esophageal Cancer with Preoperative Chemotherapy. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S1380-7. doi: 10.1245/s10434-015-4531-2. Epub 2015 May 5. PMID 25940570
- [Background] Oliver J, Garcia-Aranda M, Chaves P, Alba E, Cobo-Dols M, Onieva JL, Barragan I. Emerging noninvasive methylation biomarkers of cancer prognosis and drug response prediction. Semin Cancer Biol. 2022 Aug;83:584-595. doi: 10.1016/j.semcancer.2021.03.012. Epub 2021 Mar 20. PMID 33757849
- [Background] Komoto S, Noma K, Kato T, Kobayashi T, Nishiwaki N, Narusaka T, Sato H, Katsura Y, Kashima H, Kikuchi S, Ohara T, Tazawa H, Fujiwara T. Conventional Cancer Therapies Can Accelerate Malignant Potential of Cancer Cells by Activating Cancer-Associated Fibroblasts in Esophageal Cancer Models. Cancers (Basel). 2023 May 30;15(11):2971. doi: 10.3390/cancers15112971. PMID 37296933
- [Background] Jeong DY, Lee KS, Choi JY, Chung MJ, Min YW, Kim HK, Zo JI, Shim YM, Sun JM. Surgically Resected Esophageal Squamous Cell Carcinoma: Patient Survival and Clinicopathological Prognostic Factors. Sci Rep. 2020 Mar 19;10(1):5077. doi: 10.1038/s41598-020-62028-5. PMID 32193500
- [Background] Cao W, Lee H, Wu W, Zaman A, McCorkle S, Yan M, Chen J, Xing Q, Sinnott-Armstrong N, Xu H, Sailani MR, Tang W, Cui Y, Liu J, Guan H, Lv P, Sun X, Sun L, Han P, Lou Y, Chang J, Wang J, Gao Y, Guo J, Schenk G, Shain AH, Biddle FG, Collisson E, Snyder M, Bivona TG. Multi-faceted epigenetic dysregulation of gene expression promotes esophageal squamous cell carcinoma. Nat Commun. 2020 Jul 22;11(1):3675. doi: 10.1038/s41467-020-17227-z. PMID 32699215
- [Background] Liu Z, Zhao Y, Kong P, Liu Y, Huang J, Xu E, Wei W, Li G, Cheng X, Xue L, Li Y, Chen H, Wei S, Sun R, Cui H, Meng Y, Liu M, Li Y, Feng R, Yu X, Zhu R, Wu Y, Li L, Yang B, Ma Y, Wang J, Zhu W, Deng D, Xi Y, Wang F, Li H, Guo S, Zhuang X, Wang X, Jiao Y, Cui Y, Zhan Q. Integrated multi-omics profiling yields a clinically relevant molecular classification for esophageal squamous cell carcinoma. Cancer Cell. 2023 Jan 9;41(1):181-195.e9. doi: 10.1016/j.ccell.2022.12.004. Epub 2022 Dec 29. PMID 36584672